CLINICAL TRIAL: NCT01295671
Title: Sugar Sweetened Beverages And Cardiovascular Disease Risk
Brief Title: Beverages and Societal Health
Acronym: BASH III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, David S. Ludwig, MD, PhD, Director, Obesity Prevention Center, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-06-0242
Record Dates: First submitted 2011-02-11; First posted 2011-02-14 (Estimated); Results first posted 2018-03-27 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-02

CONDITIONS: Cardiovascular Disease, Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sugar-Sweetened Beverages (Active Comparator): Provision of beverages: Sugar-sweetened beverages
  Interventions: Behavioral: Provision of beverages
- Artificially-sweetened Beverages (Experimental): Provision of beverages: Artificially-sweetened beverages
  Interventions: Behavioral: Provision of beverages
- Unsweetened Beverages (Experimental): Provision of beverages: Unsweetened beverages
  Interventions: Behavioral: Provision of beverages

INTERVENTIONS:
Behavioral: Provision of beverages — Home delivery of specified beverage type

SUMMARY:
The overall aim of the study is to compare the effects of three types of beverages - sugar-sweetened (SSB), artificially sweetened (ASB), and unsweetened (USB) - on cardiovascular disease (CVD) risk factors and body weight among young adults.

DETAILED DESCRIPTION:
Consumption of sugar sweetened beverages (SSB) has been linked to obesity and, independent of body weight, risk for diabetes and cardiovascular disease. With rising public health awareness of these potential adverse effects, consumption of artificially sweetened beverages (ASB) has increased dramatically. These low-calorie products are marketed as "diet," with the implication that they promote weight loss and improved health. However, there are no long-term experimental studies of ASB and body weight or any other health outcome. Several recent prospective observational studies have linked intake of ASB to increased risk of the metabolic syndrome, type 2 diabetes, and obesity. In the proposed clinical trial, 270 young adults who habitually consume SSB will be randomly assigned to one of three groups: 1) to continue consuming habitual levels of SSB; 2) to substitute ASB for SSB; or 3) to substitute unsweetened beverages for SSB. Each group will receive home delivery of the targeted beverage for 1 year, using methods that build upon previous successful work. Careful attention will be given to assuring treatment fidelity, equivalence of treatment intensity, and avoidance of experimental confounders. The primary study endpoint will be the ratio of serum triglyceride to HDL-cholesterol concentrations. Secondary endpoints will include changes in other cardiovascular disease risk factors, body weight, dietary quality, and taste preferences.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 40 years
* Consumption of at least 12 fluid ounces of sugar-sweetened beverage per day
* Willingness to consume types of beverages consistent with group assignment
* Body mass index (BMI) ranging from 18.5 - 40 kg/m2, and body weight ≤275 pounds
* Access to a working telephone or cell phone

Exclusion Criteria:

* Intention to move away from the greater Boston area during the projected period of study enrollment (i.e., 1 year post-randomization)
* Plans to be away from home for 5 weeks or longer during the study period (e.g., moving away from the greater Boston area during the summer)
* Physician diagnosis of a major medical illness, eating disorder, or phenylketonuria (PKU)
* Chronic use of any medication that may affect one or more study endpoints
* Impaired fasting glucose (IFG, fasting blood glucose ≥110 mg/dL)
* Current moderate or heavy smoker (>10 cigarettes per day)
* Another member of the family (i.e., first degree relative) or household participating in the study If female,
* Pregnant in the past 12 months or planning to become pregnant during the study period
* Lactating in the preceding 3 months
* Change in birth control medication in previous 3 months or plans to change during the study period

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 203 (Actual)
Dates: Start 2011-02; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ebbeling CB, Feldman HA, Osganian SK, Chomitz VR, Ellenbogen SJ, Ludwig DS. Effects of decreasing sugar-sweetened beverage consumption on body weight in adolescents: a randomized, controlled pilot study. Pediatrics. 2006 Mar;117(3):673-80. doi: 10.1542/peds.2005-0983. PMID 16510646
- [Background] Ebbeling CB, Feldman HA, Chomitz VR, Antonelli TA, Gortmaker SL, Osganian SK, Ludwig DS. A randomized trial of sugar-sweetened beverages and adolescent body weight. N Engl J Med. 2012 Oct 11;367(15):1407-16. doi: 10.1056/NEJMoa1203388. Epub 2012 Sep 21. PMID 22998339
- [Derived] Ebbeling CB, Feldman HA, Steltz SK, Quinn NL, Robinson LM, Ludwig DS. Effects of Sugar-Sweetened, Artificially Sweetened, and Unsweetened Beverages on Cardiometabolic Risk Factors, Body Composition, and Sweet Taste Preference: A Randomized Controlled Trial. J Am Heart Assoc. 2020 Aug 4;9(15):e015668. doi: 10.1161/JAHA.119.015668. Epub 2020 Jul 22. PMID 32696704

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Boston metro area via multiple recruitment methods (i.e., print media, social media) from February 2011 through October 2014.
Pre-assignment Details: 3607 participants were initially telephone screened; 1462 were eligible after telephone screening; 407 were eligible after an Informational Visit; 222 provided informed consent; 19 withdrew or were found ineligible prior to completing baseline assessments. 203 participants completed baseline assessments and were randomized.
Period: Overall Study
Arm/Group | Sugar-Sweetened Beverages | Artificially-sweetened Beverages | Unsweetened Beverages
Started | 67 | 67 | 69
Completed | 60 | 60 | 66
Not Completed | 7 | 7 | 3
Not completed — Lost to Follow-up | 4 | 6 | 3
Not completed — Withdrawal by Subject | 3 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sugar-Sweetened Beverages: Sugar-sweetened beverages
  Provision of beverages: Home delivery of specified beverage type
- Artificially-Sweetened Beverages: Artificially-sweetened beverages
  Provision of beverages: Home delivery of specified beverage type
- Unsweetened Beverages: Unsweetened beverages
  Provision of beverages: Home delivery of specified beverage type
- Total: Total of all reporting groups
Arm/Group | Sugar-Sweetened Beverages | Artificially-Sweetened Beverages | Unsweetened Beverages | Total
Number analyzed (Participants) | 67 | 67 | 69 | 203
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 67 | 67 | 69 | 203
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.9 (5.1) | 26.7 (5.7) | 28.0 (6.0) | 26.9 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 40 | 41 | 108
  Male | 40 | 27 | 28 | 95
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 67 | 67 | 69 | 203
Ratio of Serum Triglyceride to HDL-cholesterol Concentration (TG:HDLC) [Mean (Inter-Quartile Range); unit: ratio of Triglycerides-to-HDL] | 1.37 [0.87 to 2.16] | 1.30 [0.78 to 1.98] | 1.51 [1.08 to 2.51] | 1.37 [0.90 to 2.17]
LDL-C [Mean (Standard Deviation); unit: mg/dL] | 100 (27) | 102 (28) | 110 (33) | 104 (30)
hsCRP [Median (Inter-Quartile Range); unit: mg/L] | 0.62 [0.32 to 1.84] | 0.77 [0.34 to 2.30] | 0.73 [0.43 to 1.38] | 0.69 [0.34 to 2.08]
Fibrinogen [Mean (Standard Deviation); unit: mg/dL] | 241 (64) | 241 (74) | 250 (71) | 244 (70)
Uric Acid [Mean (Standard Deviation); unit: mg/dL] | 5.3 (1.3) | 5.2 (1.4) | 5.3 (1.5) | 5.3 (1.4)
ALT [Median (Inter-Quartile Range); unit: U/L] | 14 [12 to 21] | 18 [13 to 27] | 16 [13 to 22] | 16 [13 to 22]
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 108 (9) | 109 (13) | 106 (10) | 108 (11)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 67 (8) | 67 (8) | 68 (7) | 67 (8)
Body Weight [Mean (Standard Deviation); unit: kg] | 75.5 (15.6) | 76.8 (16.7) | 77.5 (16.1) | 76.6 (16.1)
Diet Quality: Sugar-Sweetened Beverage Consumption [Mean (Standard Deviation); unit: Servings per day] | 1.4 (1.1) | 1.5 (1.4) | 1.8 (1.3) | 1.6 (1.3)
Preference for sweet taste [Median (Inter-Quartile Range); unit: Sample number] — We evaluated preference for sweet taste using ten solutions ranging in sucrose concentration (%m/v) from 0% (sample 1) to 18% (sample 10). After tasting each solution, participant reported the sample number corresponding to his or her overall favorite.
  Sample number | 6 [5 to 7] | 6 [5 to 8] | 7 [5 to 7] | 6 [5 to 8]

OUTCOME MEASURES:

1. Primary Outcome: Ratio of Serum Triglyceride to HDL-cholesterol Concentration (TG:HDLC)
Time Frame: 12 Month
Measure: Median (Inter-Quartile Range); unit: ratio of Triglycerides-to-HDL
Arm/Group | Sugar-Sweetened Beverages | Artificially-sweetened Beverages | Unsweetened Beverages
Number analyzed (Participants) | 60 | 60 | 66
ratio of Triglycerides-to-HDL | 1.46 [0.98 to 2.19] | 1.19 [0.86 to 1.87] | 1.45 [0.99 to 2.31]

2. Secondary Outcome: LDL-C
Description: LDL-C
Time Frame: 12 Month
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Sugar-Sweetened Beverages | Artificially-sweetened Beverages | Unsweetened Beverages
Number analyzed (Participants) | 60 | 60 | 66
mg/dL | 103 (31) | 104 (30) | 109 (29)

3. Secondary Outcome: hsCRP
Description: hsCRP
Time Frame: 12 Month
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Sugar-Sweetened Beverages | Artificially-sweetened Beverages | Unsweetened Beverages
Number analyzed (Participants) | 60 | 60 | 66
mg/L | 0.86 [0.39 to 1.80] | 0.64 [0.39 to 1.81] | 0.85 [0.39 to 1.76]

4. Secondary Outcome: Fibrinogen
Description: Fibrinogen
Time Frame: 12 Month
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Sugar-Sweetened Beverages | Artificially-sweetened Beverages | Unsweetened Beverages
Number analyzed (Participants) | 60 | 60 | 66
mg/dL | 244 (49) | 248 (62) | 236 (73)

5. Secondary Outcome: Uric Acid
Description: Uric Acid
Time Frame: 12 Month
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Sugar-Sweetened Beverages | Artificially-sweetened Beverages | Unsweetened Beverages
Number analyzed (Participants) | 60 | 60 | 66
mg/dL | 5.2 (1.3) | 5.1 (1.4) | 5.4 (1.5)

6. Secondary Outcome: ALT
Description: ALT
Time Frame: 12 Month
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Sugar-Sweetened Beverages | Artificially-sweetened Beverages | Unsweetened Beverages
Number analyzed (Participants) | 60 | 60 | 66
U/L | 16 [12 to 21] | 16 [13 to 23] | 17 [11 to 26]

7. Secondary Outcome: Systolic Blood Pressure
Description: Systolic Blood Pressure
Time Frame: 12 Month
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sugar-Sweetened Beverages | Artificially-sweetened Beverages | Unsweetened Beverages
Number analyzed (Participants) | 60 | 60 | 66
mmHg | 109 (10) | 107 (11) | 106 (9)

8. Secondary Outcome: Diastolic Blood Pressure
Description: Diastolic Blood Pressure
Time Frame: 12 Month
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sugar-Sweetened Beverages | Artificially-sweetened Beverages | Unsweetened Beverages
Number analyzed (Participants) | 60 | 60 | 66
mmHg | 68 (9) | 67 (8) | 67 (8)

9. Secondary Outcome: Body Weight
Description: Body Weight
Time Frame: 12 Month
Population: Data missing for 1 subject in ASB group.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Sugar-Sweetened Beverages | Artificially-sweetened Beverages | Unsweetened Beverages
Number analyzed (Participants) | 60 | 59 | 66
kg | 78.0 (17.4) | 76.8 (17.2) | 78.3 (17.1)

10. Secondary Outcome: Diet Quality: Sugar-Sweetened Beverage Consumption
Description: Diet Quality: Sugar-Sweetened Beverage Consumption - servings per day
Time Frame: 12 Month
Population: Data missing for 1 subject in USB group.
Measure: Mean (Standard Deviation); unit: Servings per day
Arm/Group | Sugar-Sweetened Beverages | Artificially-sweetened Beverages | Unsweetened Beverages
Number analyzed (Participants) | 60 | 60 | 65
Servings per day | 2.5 (1.8) | 0.1 (0.3) | 0.2 (2.5)

11. Secondary Outcome: Preference for Sweet Taste
Description: We evaluated preference for sweet taste using ten solutions ranging in sucrose concentration (%m/v) from 0% (sample 1) to 18% (sample 10). After tasting each solution, participant reported the sample number corresponding to his or her overall favorite.
Time Frame: 12 Month
Population: Data missing for 1 subject in SSB group.
Measure: Median (Inter-Quartile Range); unit: Sample number
Arm/Group | Sugar-Sweetened Beverages | Artificially-sweetened Beverages | Unsweetened Beverages
Number analyzed (Participants) | 59 | 60 | 66
Sample number | 6 [5 to 7] | 6 [4.5 to 7] | 5 [4 to 6]

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Group 1: Sugar-sweetened beverages
  Provision of beverages: Home delivery of specified beverage type
- Group 2: Artificially-sweetened beverages
  Provision of beverages: Home delivery of specified beverage type
- Group 3: Unsweetened beverages
  Provision of beverages: Home delivery of specified beverage type
Arm/Group | Group 1 | Group 2 | Group 3
Serious Adverse Events (participants affected / at risk) | 2/67 | 1/67 | 0/69
Other Adverse Events (participants affected / at risk) | 0/67 | 0/67 | 0/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=67) | Group 2 (N=67) | Group 3 (N=69)
Body Aches (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Hospitalized for pain management of a severely pulled muscle in chest.
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — Hospitalized for asthma
Headaches and mood swings due to toothache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Severe headaches and mood swings due to toothache

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No